CLINICAL TRIAL: NCT01192893
Title: Role of Oxytocin in Post-menopausal Osteoporosis: Evaluation on the Population of the OPUS Cohort
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 10-PP-07
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — OPUS is a prospective study of postmenopausal women recruited in the general population between April 1999 and April 2001 from five European centers (Aberdeen (UK), Berlin (Germany), Kiel (Germany), Paris (Hôpital Cochin, France), and Sheffield (UK)). Investigations were approved at each institution according to the Declaration of Helsinki. Written consent was obtained from all subjects. Each center recruited approximately 500 postmenopausal women comprising 100 individuals in each 5-yr age band between 55 and 79. Ninety-nine percent of subjects were of white ethnicity.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OPUS: OPUS is a prospective study of postmenopausal women recruited in the general population between April 1999 and April 2001 from five European centers (Aberdeen (UK), Berlin (Germany), Kiel (Germany), Paris (Hospital Cochin, France), and Sheffield (UK)). Investigations were approved at each institution according to the Declaration of Helsinki. Written consent was obtained from all subjects. Each center recruited approximately 500 postmenopausal women comprising 100 individuals in each 5-yr age band between 55 and 79. Ninety-nine percent of subjects were of white ethnicity.

SUMMARY:
Oxytocin is a neurohypophysial hormone involved in several central and peripheral functions including parturition, milk let-down reflex and social behaviour. In vitro and animals studies have shown growing evidence that oxytocin plays a role in bone remodeling and osteoporosis. The investigators have previously show in a small sample of post-menopausal women with severe osteoporosis (n=20) compare to healthy control (n=16) that oxytocin serum level is significantly decreased, independently of leptin and estradiol, that are known to modulate oxytocin secretion. Thus, oxytocin appears as a new interesting factor in the osteoporosis pathophysiology. The aim of the present study is to confirm the relationships between bone status, evaluated by bone mineral density and prevalent fragility fractures, body composition and oxytocin serum levels on a large population. The investigators will also determine if the relationship between bone mineral density and oxytocin is independent of estradiol and leptin in this population and evaluate the relationships between oxytocin serum level and co-morbidities such as cardiovascular diseases, depression and dementia. Theses analysis will be done on the serum already available of 1000 women of the international OPUS cohort. Bone mineral density, body composition analysis by Dual energy X-ray Absorptiometry (DXA), estradiol and clinical data are already available. The investigators will select women, aged from 55 to 79 y at the time of inclusion.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal women,
* able to undergo bone density,
* without cognitive limitation,
* Age at the time of inclusion: 55 -79y,
* Written consent.

Exclusion Criteria:

* Individuals were excluded because of inability to undergo bone densitometry or perform specified investigations or because of cognitive limitations

Ages: 55 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OPUS is a prospective study of postmenopausal women recruited in the general population between April 1999 and April 2001 from five European centers (Aberdeen (UK), Berlin (Germany), Kiel (Germany), Paris (Hôpital Cochin, France), and Sheffield (UK)). Investigations were approved at each institution according to the Declaration of Helsinki. Written consent was obtained from all subjects. Each center recruited approximately 500 postmenopausal women comprising 100 individuals in each 5-yr age band between 55 and 79. Ninety-nine percent of subjects were of white ethnicity.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
oxytocin serum levels | at time = 0
  oxytocin serum levels, measured by radio-immuno assay, at the spine and the hip in post-menopausal women
bone mineral density | at time = 0
  bone mineral density, measured by dual X ray absorptiometry at the spine and the hip in post-menopausal women

SECONDARY OUTCOMES:
Estradiol serum level | at time = 0
  Estradiol serum level, body composition (lean mass and fat mass), measured by dual X ray absorptiometry, clinical data (age, age of menopause, previous family history of hip fracture, personal prevalent osteoporotic fractures, prevalent cardiovascular disease, depression and dementia)
leptin serum level | at time = 0
  Leptinserum level, body composition (lean mass and fat mass), measured by dual X ray absorptiometry, clinical data (age, age of menopause, previous family history of hip fracture, personal prevalent osteoporotic fractures, prevalent cardiovascular disease, depression and dementia)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Archet 1, Nice, France

REFERENCES:
- [Derived] Breuil V, Fontas E, Chapurlat R, Panaia-Ferrari P, Yahia HB, Faure S, Euller-Ziegler L, Amri EZ, Szulc P. Oxytocin and bone status in men: analysis of the MINOS cohort. Osteoporos Int. 2015 Dec;26(12):2877-82. doi: 10.1007/s00198-015-3201-3. Epub 2015 Jun 25. PMID 26109496
- [Derived] Breuil V, Panaia-Ferrari P, Fontas E, Roux C, Kolta S, Eastell R, Ben Yahia H, Faure S, Gossiel F, Benhamou CL, Euller-Ziegler L, Amri EZ. Oxytocin, a new determinant of bone mineral density in post-menopausal women: analysis of the OPUS cohort. J Clin Endocrinol Metab. 2014 Apr;99(4):E634-41. doi: 10.1210/jc.2013-4126. Epub 2014 Jan 21. PMID 24446658